CLINICAL TRIAL: NCT07135973
Title: A Multi-center, Single-arm Phase IV Clinical Trial to Evaluate the Safety of Belumosudil in Indian Participants, 12 Years and Above, With Chronic Graft-versus-host Disease (cGVHD)
Brief Title: A Study to Investigate Safety of Belumosudil in Participants Aged 12 Years and Above, With Chronic Graft-versus-host Disease (cGVHD)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LPS18471
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — belumosudil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- belumosudil (Experimental): 200 mg taken orally once daily with food for 24 weeks
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil — Pharmaceutical form:Tablet-Route of administration:Oral
  Other Names: SAR445761; Rezurock

SUMMARY:
This is an interventional phase IV clinical study which is single-arm study for assessing the safety of belumosudil in Indian patients who are12 years and older.

Study details include:

* The study duration will be up to 12 months per participant.
* The treatment duration will be up to 24 weeks.
* The number of visits will be 7.

ELIGIBILITY:
Inclusion Criteria: Male or female patients at least 12 years of age inclusive, at the time of signing the informed consent Participants who had an allogeneic hematopoietic cell transplantation (HCT) Previously received at least 2 prior lines of systemic therapy for cGVHD Received glucocorticoid therapy with a stable dose over the 2 weeks prior to screening Had persistent cGVHD manifestations and systemic therapy was indicated Karnofsky (if aged ≥ 16 years)/Lansky (if aged <16 years) Performance Score of ≥ 60

Capable of giving signed informed consent as described in the protocol Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

Absolute neutrophil count ≤1.5 X 109/L Platelet count ≤ 50 X 109/L Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 3 X upper limit of normal (ULN) (>5 × ULN if due to cGVHD) Total bilirubin ≥ 1.5 X ULN Glomerular filtration rate (GFR) ≤ 30 mL/min/1.73m3 Positive hepatitis B surface antigen, or hepatitis C antibody or HIV antibody at screening FEV1 ≤39% or has lung score of 3

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-11-28 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-03-17 (Estimated)

PRIMARY OUTCOMES:
Drug related Grade ≥ 3 treatment emergent adverse events (TEAE) | From baseline to 24 weeks
  Drug related Grade ≥ 3 treatment emergent adverse events (TEAE) during the treatment period (24 weeks)

SECONDARY OUTCOMES:
Best overall Response (BoR) | Baseline to end of study i.e. 12 months
  Best overall Response (BoR), defined as the proportion of patients who achieved complete response (CR) or partial response (PR) according to the NIH Consensus Criteria.
Duration of Response (DOR) | Baseline to end of study i.e. 12 months
  Duration of Response (DOR) calculated from time of initial PR or CR until documented progression, death, or new systemic therapy.
Time to Response (TTR) | Baseline to end of study i.e. 12 months
Response by organ system (including GSR) | Baseline to end of study i.e. 12 months
Time taken for New Treatment (TTNT) or death | Baseline to end of study i.e. 12 months
Failure-free survival (FFS) | Baseline to end of study i.e. 12 months
Overall survival (OS) | Baseline to end of study i.e. 12 months
Change in Corticosteroid dose. | Baseline to end of study i.e. 12 months
Change in CNI dose | Baseline to end of study i.e. 12 months
Symptomatic improvement from baseline during treatment based on modified Lee Symptom Scale | Baseline to end of study i.e. 12 months
  defined as a ≥7-point reduction from baseline in total symptom score on a scale of 0 to 100 which measures the symptoms of chronic GVHD, with higher scores indicating worse symptoms
Pulmonary Function Test (PFT) | Baseline to end of study i.e. 12 months
  Total lung capacity, Residual volume, Forced expiratory volume, Tidal volume
Number of participants with treatment-emergent adverse events [TEAEs], serious TEAEs, and adverse events of special interest (AESIs) | Baseline to end of study i.e. 12 months

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org